CLINICAL TRIAL: NCT03697135
Title: A Respondent Driven Sampling Study to Identify the Hidden Population of Former Intravenous Drug Users With Hepatitis C Infection Who Are no Longer in Contact With Services. "Ask a Friend"
Brief Title: Ask a Friend to Take a Test for Hepatitis C Infection
Status: Completed | Type: Observational
Sponsor: NHS Tayside (Other Government)
Collaborators: University of Dundee (Other)
Responsible Party: Principal Investigator, Andrew Radley, Consultant in Public Health Pharmacy, NHS Tayside
Other Study IDs: 2016GA02
Record Dates: First submitted 2018-03-23; First posted 2018-10-05 (Actual); Last update posted 2020-08-04 (Actual); Status verified 2020-07

CONDITIONS: Hepatitis C
MeSH Terms: conditions — Hepatitis C

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Seed Contacts: Initial participants who will invite previous injecting contacts to take a hepatitis C test using a respondent driven sampling method
  Interventions: Behavioral: Respondent Driven Sampling
- Initial Nominations for Testing: Contacts of initial participants who consent to be tested and enrol in the study using a respondent driven sampling method
  Interventions: Behavioral: Respondent Driven Sampling
- Second Level Nominations for testing: Contacts of wave one participants who consent to be tested and enrol in the study using a respondent driven sampling method
  Interventions: Behavioral: Respondent Driven Sampling

INTERVENTIONS:
Behavioral: Respondent Driven Sampling — Participants are asked to invite contacts that they previously injected with to take a test for hepatitis C

SUMMARY:
This exploratory study will carry out a respondent-driven sampling exercise, where participants will identify their previous injecting partners and contact these individuals to invite them to take an Hepatitis C test. The data from participants about their injecting network will be used to construct a social network map (egonet) of the interlinking injecting networks. The numbers of individuals identified in the injecting networks will be used to estimate the size of the injecting population in Dundee. Participants will be interviewed to find out how they felt about the processes used.

DETAILED DESCRIPTION:
Initial seed participants (25 individuals) will be identified from local support organisations who work with drug users, by members of the research team. Members of the research team will identify seeds from the Cairn Centre initially and sequentially visit partner organisations as the study proceeds. Seed participants will be current or former injecting drug users who are in contact with services. Seed participants will be provided with the study information sheet (PIS, participant information sheet) and asked to provide consent to take part in the study, according to standard practice. All members of the research team are trained in study procedures and Good Clinical Practice Seed participants will be requested to identify members of their previous injecting network by providing general information about these individuals to create a pseudo-identity. They may be assisted in doing this by the use of a mapping tool. The researchers will collect a standard dataset: Given name; approximate age; approximate area of town/city (if known); Ethnicity; Strength of tie (How often they injected with this person - Likert scale, year first and last injected with). The pseudo-identities created by the seeds will be insufficient to identify an actual person, but will enable the seed participant to focus on who they might like to contact. The actual identities of the person they contact will only be known to the researchers when this person presents for testing and consents to participation.

Advice will be given to the seed participants about sensitively approaching individuals who they used to inject with and about how people who are approached by them can access HCV testing. The data from identified contacts will be recorded onto an Excel Spreadsheet held on a password-protected computer within a locked office at the University of Dundee. These data will be utilised to construct an egomap using a computer programme designed for this purpose such as "Egonet". However it should be noted that the identified contacts are "pseudo identities" since the details do not correspond to a real person until they come forward for testing and can be linked to a CHI number.

Seed participants will have the study coupon system explained to them, which they will use to invite injecting partners to take an HCV test. Each study coupon will contain a unique reference number that links it to the individual who gave the former IDU the invitation. The participants will be handed sufficient coupons to cover the number of alters identified by them, up to a maximum of 5 coupons at one time. The seed participants will be issued with study information cards and study coupons to enable them to invite their contacts to present for an HCV test. The former drug users identified by seeds represent wave 1 of the respondent-driven sample. The respondent driven sampling will be managed with standard software (RDSAT). If seeds only identify contacts known to services, then this will be recorded and the participant's social network logged.

Seed participants will be contacted weekly by phone or when they are visiting the Cairn Centre for up to 4 weeks, by a designated member of the research team to ask about progress in contacting social network contacts. The contact will be recorded on a log sheet that will enable a summary of the conversation to be recorded The study will initially offer Dried Blood Spot Testing (DBST) through the Cairn Centre in Dundee, where the study methods will be first piloted. Individuals who wish to be tested will contact the Cairn Centre using the telephone number included on the coupon and make an arrangement to be tested. All testing will be done according to the standard operating procedures and guidance prepared by the Sexual Health and Blood Borne Virus Managed Care Network.

As the study proceeds, additional sites will be visited by the research team and additional seeds identified and invited to participate if required. These additional sites are already in use by the intended participant groups as community hubs and community pharmacies in Dundee at Lochee, Hilltown, Albert Street and Menzieshill. At this stage, potential participants may be approached by the care team (community/pharmacy) only who will introduce the research team to potential participants When the potential wave 1 study participant (who is a contact identified by the seed participant) contacts the Cairn Centre about a DBST, all relevant details to enable their clinical care will be recorded by the member of the specialist nurse, who works in the Cairn Centre, to enable the results of the test to be communicated to the participant and advice on any future care and treatment provided. The information collected will be sufficient to enable a CHI number to be identified. The CHI number is an essential requirement to ensure that all participants who are tested can be informed of the test result and can access ongoing referral and treatment as appropriate. The processing of results and documentation in the clinical record will be undertaken by a research nurse attached to the HCV clinical team. The participant will be provided with information about the HCV test and its meaning and offered referral for treatment as NHS standard of care. In addition and making it clear this is an additional option the nurse will give a PIS, to advise them about the opportunity to join the study. Caldicott approvals will be gained for all appropriate data that will be collected At least 24 hours after they have received study information they will be asked if they will consent to participate in the study and then visit the Cairn Centre for a test. Wave 1 participants will be invited to provide standard information about people that they injected with, as described above, to enable an egomap to be constructed. The participant will be supported to complete a standard form containing the minimum dataset required to construct the egomap. The Standard dataset is: Name; approximate age; area of town/city; Ethnicity; Strength of tie (How often they injected with this person - Likert scale). Specialist nurses from the clinical team who work at the Cairn Centre will talk to Seeds about sensitively approaching individuals who they have discussed who they used to inject with and about how people who are approached can access HCV testing. The information collected will be used to identify how many potential contacts the participant has knowledge of and compared to the actual recruitment and to ascertain the relationships between one injecting network and an adjacent network.

The people handed coupons by the Wave 1 participants will constitute Wave 2 participants. When the wave 2 participant present for HCV testing, the person testing them will follow the same procedure as outlined above so that the participant can be advised of their test result and be referred for on-going care and treatment if required. The wave 2 participants will receive the same training and guidance as the wave one participants received. Study procedures regarding inclusion, exclusion and consent will be identical for each Wave.

ELIGIBILITY:
Inclusion criteria for the study are as follows:

* Previous or current history of injecting drug use
* Able to provide informed consent
* Willing to identify previous injecting partners (people they have injected with)
* Willing to undergo training on approaching previous injecting partners according to the study proceduresWilling to contact previous injecting partners according to the study proceduresAged 18 and over

Exclusion criteria for the study are as follows:

* No previous history of injecting drug use
* Not willing to provide informed consentNot willing to participate in the procedures required in the study protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Injecting partners of people who use drugs
Sampling Method: Non-Probability Sample
Enrollment: 51 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2019-12-30 (Actual); Study Completion 2019-12-30 (Actual)

PRIMARY OUTCOMES:
Hepatitis C test | baseline
  Number of participants consenting to a Hepatitis C test by Dried Blood Spot

SECONDARY OUTCOMES:
Process evaluation | baseline
  Qualitative interview with each participant using discussion guide agreed by ethics

CONTACTS AND LOCATIONS:
Overall Officials: John Dillon, MD, Study Director — University of Dundee
Locations (1):
- Ninewells Hospital, Dundee, Tayside, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided
Anonymised social network structures of a hepatitis C injecting network

REFERENCES:
- [Background] Abdul-Quader AS, Heckathorn DD, McKnight C, Bramson H, Nemeth C, Sabin K, Gallagher K, Des Jarlais DC. Effectiveness of respondent-driven sampling for recruiting drug users in New York City: findings from a pilot study. J Urban Health. 2006 May;83(3):459-76. doi: 10.1007/s11524-006-9052-7. PMID 16739048
- [Background] Heckathorn DD, Semaan S, Broadhead RS, Hughes JJ. Extensions of respondent-driven sampling: a new approach to the study of injection drug users aged 18-25. AIDS and Behavior. 2002;6(1):55-67.
- [Derived] Donaldson SR, Radley A, Dillon JF. Identifying the Hidden Population: Former Intravenous Drug Users Who Are No Longer in Contact with Services. "Ask a Friend". Diagnostics (Basel). 2021 Jan 25;11(2):170. doi: 10.3390/diagnostics11020170. PMID 33504077